CLINICAL TRIAL: NCT05603195
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single-Center Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single Ascending Doses of REGN7508, a Monoclonal Antibody Against Factor XI, in Healthy Adult Subjects
Brief Title: A Trial to Learn if Single Ascending Intravenous (IV) Doses of REGN7508 Are Safe and Well Tolerated, and How it Works in the Body of Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R7508-HV-21102; 2022-002001-20 (EudraCT Number)
Record Dates: First submitted 2022-10-27; First posted 2022-11-02 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Healthy Volunteer
Keywords: Thrombotic disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (10):
- Cohort 1 Lowest IV Dose (Experimental): Randomized 3:1
  Interventions: Drug: REGN7508 (IV); Drug: Matching Placebo (IV)
- Cohort 2 Low IV Dose (Experimental): Randomized 3:1
  Interventions: Drug: REGN7508 (IV); Drug: Matching Placebo (IV)
- Cohort 3 Mid IV Dose (Experimental): Randomized 3:1
  Interventions: Drug: REGN7508 (IV); Drug: Matching Placebo (IV)
- Cohort 4 High IV Dose (Experimental): Randomized 3:1
  Interventions: Drug: REGN7508 (IV); Drug: Matching Placebo (IV)
- Cohort 5 Higher IV Dose (Experimental): Randomized 3:1
  Interventions: Drug: REGN7508 (IV); Drug: Matching Placebo (IV)
- Cohort 6 High SC Dose (Experimental): Randomized 3:1
  Interventions: Drug: REGN7508 (SC); Drug: Matching Placebo (SC)
- Cohort 7 Higher SC Dose (Experimental): Randomized 3:1
  Interventions: Drug: REGN7508 (SC); Drug: Matching Placebo (SC)
- Optional: Cohort 8 Highest IV or SC Dose (Experimental): Randomized 3:1
  Interventions: Drug: REGN7508 (IV); Drug: REGN7508 (SC); Drug: Matching Placebo (IV); Drug: Matching Placebo (SC)
- Cohort 9 High SC Dose (Experimental): Randomized 3:1
  Interventions: Drug: REGN7508 (SC); Drug: Matching Placebo (SC)
- Optional: Cohort 10 Highest SC Dose (Experimental): Randomized 3:1
  Interventions: Drug: REGN7508 (SC); Drug: Matching Placebo (SC)

INTERVENTIONS:
Drug: REGN7508 (IV) — Administered sequential, ascending single intravenous (IV) dose
  Arms: Cohort 1 Lowest IV Dose; Cohort 2 Low IV Dose; Cohort 3 Mid IV Dose; Cohort 4 High IV Dose; Cohort 5 Higher IV Dose; Optional: Cohort 8 Highest IV or SC Dose
Drug: REGN7508 (SC) — Administered sequential, ascending single subcutaneous (SC) dose
  Arms: Cohort 6 High SC Dose; Cohort 7 Higher SC Dose; Cohort 9 High SC Dose; Optional: Cohort 10 Highest SC Dose; Optional: Cohort 8 Highest IV or SC Dose
Drug: Matching Placebo (IV) — Administered sequential, ascending single intravenous (IV) dose
  Arms: Cohort 1 Lowest IV Dose; Cohort 2 Low IV Dose; Cohort 3 Mid IV Dose; Cohort 4 High IV Dose; Cohort 5 Higher IV Dose; Optional: Cohort 8 Highest IV or SC Dose
Drug: Matching Placebo (SC) — Administered sequential, ascending single subcutaneous (SC) dose
  Arms: Cohort 6 High SC Dose; Cohort 7 Higher SC Dose; Cohort 9 High SC Dose; Optional: Cohort 10 Highest SC Dose; Optional: Cohort 8 Highest IV or SC Dose

SUMMARY:
This study is researching an experimental drug called REGN7508 (called "study drug"). The aim of this study is to see how safe and tolerable the study drug is in healthy participants.

This study is looking at several other research questions, including:

* What side effects may happen from taking the study drug
* How much study drug is in the blood at different times
* Whether the body makes antibodies against the study drug (which could make the drug less effective or could lead to side effects)

ELIGIBILITY:
Key Inclusion Criteria:

1. Body mass index between 18.0 and 32.5 kg/m2 (inclusive) at the screening visit
2. Judged by the investigator to be in good health based on medical history, physical examination, vital sign measurements, and echocardiograms (ECGs) performed at screening and/or prior to administration of initial dose of study drug
3. Participant is in good health based on laboratory safety testing obtained at the screening visit and/or prior to administration of initial dose of study drug
4. Normal activated partial thromboplastin time (aPTT), normal prothrombin time (PT), and normal platelet counts at screening period and at the day -1 visit as defined by the local laboratory
5. Hemoglobin value ≥11.0 g/dL for females and ≥12.9 g/dL for males at the screening and day 1 visits

Key Exclusion Criteria:

1. History of any major surgical procedure or clinically significant physical trauma, in the opinion of the investigator, that may pose a risk to the participant by study participation
2. Whole blood donation within the previous 56 days or plasma donation within the previous 7 days prior to the screening visit
3. History of clinically significant cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, psychiatric, neurological, or dermatologic disease, as assessed by the investigator, that may confound the results of the study or poses an additional risk to the participant by study participation, as defined in the protocol
4. Estimated glomerular filtration rate (eGFR) of <60 mL/min/1.73m2 at screening
5. Current smoker or former smoker, including e-cigarettes, who stopped smoking within 12 months prior to the screening visit
6. Confirmed positive drug test result at the screening visit and/or prior to randomization or a history of drug abuse within a year prior to the screening visit
7. History of alcohol abuse within the last 2 years prior to the day 1 visit
8. Any malignancy, except for nonmelanoma skin cancer or cervical/anus in situ, that have been resected with no evidence of metastatic disease for 3 years prior to the screening visit
9. History of significant multiple and/or severe allergies (eg, latex gloves) or has had an anaphylactic reaction to prescription or nonprescription drugs or food

NOTE: Other Protocol Defined Inclusion / Exclusion Criteria Apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2023-01-12 (Actual); Primary Completion 2024-09-17 (Actual); Study Completion 2024-09-17 (Actual)

PRIMARY OUTCOMES:
Incidences of treatment-emergent adverse events (TEAE) | Up to 36 days
  Treatment-emergent adverse events are defined as those that are not present at baseline or represent the exacerbation of a pre-existing condition during the on-treatment period.
Severity of TEAE | Up to 36 days
  Treatment-emergent adverse events are defined as those that are not present at baseline or represent the exacerbation of a pre-existing condition during the on-treatment period.

SECONDARY OUTCOMES:
Change from baseline in activated partial thromboplastin time (aPTT) | Up to 36 days
Change from baseline in prothrombin time (PT) | Up to 36 days
Concentrations of total REGN7508 in serum | Up to 36 days
Concentrations of functional REGN7508 in plasma | Up to 36 days
Absolute concentration and change from baseline in total Factor XI (FXI) concentrations | Up to 36 days
Absolute concentration and change from baseline in free FXI concentrations | Up to 36 days
Incidence of antidrug antibodies (ADAs) to REGN7508 over time | Up to 36 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (1):
- Labcorp Clinical Research Unit, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication, has made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry), has the legal authority to share the data, and has ensured the ability to protect participant privacy.
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/